CLINICAL TRIAL: NCT04392076
Title: The Immune and Inflammatory Profile of Patients After Image Guided Ablation of Renal Cancer With Radiofrequency Ablation (RFA)/ Microwave Ablation (MWA) vs. Cryoablation (CRYO)
Brief Title: Image Guided RFA/MWA/CRYO of RCC Biomarker Profile Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Tze Min Wah, Consultant Radiologist, University of Leeds
Other Study IDs: 124413
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Renal Cancer
Keywords: Radiofrequency ablation (RFA); Microwave ablation (MWA); Cryoablation (CRYO); Biomarker
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This is a prospective single-centre non-interventional study, collecting plasma and serum samples for immediate biomarker studies with residual samples stored for future research within an RTB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Radiofrequency Ablation (RFA) of RCC: Patients following image guided radiofrequency ablation (RFA) of renal cell carcinoma (RCC)
  Interventions: Procedure: Image Guided Ablation
- Microwave Ablation (MWA) of RCC: Patients following image guided microwave ablation (MWA) of renal cell carcinoma (RCC)
  Interventions: Procedure: Image Guided Ablation
- Cryoablation (CRYO) of RCC: Patients following image guided cryoablation (CRYO) of renal cell carcinoma (RCC)
  Interventions: Procedure: Image Guided Ablation

INTERVENTIONS:
Procedure: Image Guided Ablation — Image Guided Ablation with RFA, MWA or CRYO of Renal Cancer

SUMMARY:
Often kidney cancer is diagnosed when the tumour is small and hasn't spread. Rather than major surgery to remove the whole kidney, image-guided ablation involving heat (microwave or radiofrequency) or freezing (cryotherapy) is often used to destroy the tumour using minimal invasive technique with much less risk and discomfort. Limited evidence suggests that ablation also activates the immune system which may help in fighting the cancer. We will investigate the immune and other changes by analysing blood samples from patients before and after ablation. Understanding this will help in designing more effective new treatments combining ablation with biological therapies.

DETAILED DESCRIPTION:
Image-guided ablation therapies are increasingly being used in renal and other cancers as an alternative to major surgery, particularly in the context of small localised masses or when patients have significant co-morbidities. Published analyses now also support the effectiveness of such treatments in terms of outcomes. Tumour ablation has been reported to generate immune and inflammatory responses following tumour destruction, essentially through release of tumour antigens in effect acting as a tumour "vaccine", resulting in systemic anti-tumour responses. Such studies are still limited but indicate possibilities in terms of combination therapies with immunotherapies and synergistic effects.

In order to take this forward in renal cancer it is now critical that studies are undertaken to explore further the immunobiological and inflammatory changes associated with ablation therapies. We propose to do this using a relatively new multiplex and highly sensitive proteomic biomarker array technology which allows the profiling of circulating proteins using arrays targeted at specific disease areas or processes. We have used this platform to generate some pilot data on RCC patients undergoing ablation to show feasibility and now propose to extend this further. The main benefits to patients will be in terms of understanding how the immune and inflammatory responses are affected by ablation which ultimately may lead to the design of new more effective therapeutic strategies combining ablation with immunotherapies. Ultimately more effective combination therapies would have health economic benefits and improved quality of life with potentially lower toxicity if the doses of the biological therapies could be reduced. Some of the protein changes may also act as surrogate markers of response and guide optimal treatment administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent image guided ablation for renal cell carcinoma (RCC) with heat-based energy (RFA/MWA) or ice-based energy (CRYO)
2. No other prior treatment to RCC in either kidneys

Exclusion Criteria:

1. Patients with RCC that is not suitable for image guided ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RCC that are identified through renal cancer MDT and have agreed to undergo image guided ablation of RCC with thermal ablative technologies such as RFA, MWA or CRYO.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the immune and inflammatory response to MWA/RFA and CRYO based on plasma protein profiling using multiplex arrays and how consistent the changes are between patients and treatment type. | 15 months
  The data will be important in understanding how the immune and inflammatory responses are affected by ablation which ultimately may lead to the design of new more effective therapeutic strategies combining ablation with immunotherapies.
To analyse the profiles using biostatistical and bioinformatic tools to understand the immunopathological changes and understanding how such ablation therapies may be used in combination with immunotherapies for increased efficacy. | 15 months
  The data will be important in understanding how the immune and inflammatory responses are affected by ablation which ultimately may lead to the design of new more effective therapeutic strategies combining ablation with immunotherapies.

CONTACTS AND LOCATIONS:
Overall Officials: Tze Min Wah, PhD MBchB, Principal Investigator — Leeds Teaching Hospitals Trust
Locations (1):
- Leeds Institute of Medical Research, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided